CLINICAL TRIAL: NCT02485184
Title: TIPS Versus Endoscopic Therapy for the Prevention of Variceal Rebleeding in Cirrhotic Patients With Portal Vein Thrombosis: A Randomized Controlled Trial
Brief Title: TIPS vs Endoscopic Therapy for Variceal Rebleeding in Cirrhotic Patients With Portal Vein Thrombosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Collaborators: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Shandong Provincial Hospital (Other Government); Third Affiliated Hospital, Sun Yat-Sen University (Other); Southern Medical University, China (Other); First Affiliated Hospital of Xinjiang Medical University (Other); The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Guohong Han, Professor, Xi'an International Medical Center Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PVT-TIPS2
Record Dates: First submitted 2015-06-23; First posted 2015-06-30 (Estimated); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Portal Vein Thrombosis; Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Portasystemic Shunt, Transjugular Intrahepatic; Propranolol; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TIPS group (Active Comparator): Transjugular intrahepatic portosystemic shunt
  Interventions: Procedure: Transjugular intrahepatic portosystemic shunt
- ET & drugs groups (Active Comparator): 1. Endoscopic therapy.
  2. Non-selective beta blockers.
  3. Anticoagulation therapy.
  Interventions: Drug: Non-selective beta blockers; Procedure: Endoscopic therapy; Drug: Anticoagulation

INTERVENTIONS:
Procedure: Transjugular intrahepatic portosystemic shunt — Transjugular intrahepatic portosystemic shunt refers to an interventional radiological procedure by placing a stent between portal vein and hepatic vein. No specific device was used in the Interventional field.
  Arms: TIPS group
Drug: Non-selective beta blockers — Non-selective beta blockers are the drugs for reducing the portal pressure.
  Other Names: propranolol
  Arms: ET & drugs groups
Procedure: Endoscopic therapy — Endoscopic therapy includes the endoscopic variceal band ligation
  Arms: ET & drugs groups
Drug: Anticoagulation — Anticoagulation therapy includes heparin and warfarin.
  Other Names: warfarin
  Arms: ET & drugs groups

SUMMARY:
portal vein thrombosis may be a negative prognostic marker of variceal bleeding in liver cirrhosis. Compared with conventional endoscopic and pharmacological therapy, transjugular intrahepatic portosystemic shunt may further improve the outcomes of portal vein thrombosis in liver cirrhosis with variceal bleeding.

DETAILED DESCRIPTION:
Portal vein thrombosis may be a negative prognostic marker of variceal bleeding in liver cirrhosis. Compared with conventional endoscopic and pharmacological therapy, transjugular intrahepatic portosystemic shunt may further improve the outcomes of portal vein thrombosis in liver cirrhosis with variceal bleeding. However, the safety of transjugular intrahepatic portosystemic shunt remains uncertain in patients with portal vein thrombosis.

ELIGIBILITY:
Inclusion criteria

1. liver cirrhosis (histological or clinical);
2. Significant variceal bleeding >5 days and ≤ 42 days
3. Successful treatment of the index bleed by means of vasoactive drugs and/or endoscopic treatment
4. Portal vein thrombosis occlusion>=25% of the vessel lumen;
5. Presence of ascites
6. Child-Pugh score 8-12 at inclusion
7. Age 18 to 70 years

Exclusion criteria

1. Bleeding from isolated gastric or ectopic varices
2. Contraindications to non-selective beta blockers (chronic obstructive pulmonary disease, asthma, aortic stenosis, atrioventricular block, intermittent claudication, and psychosis)
3. Contraindications to TIPS : extensive potral vein thrombosis, fibrotic cord replacing original main portal vein; bilirubin>3.5 mg/dL, plasma creatinine>2.1 mg/dL, Child-Pugh score >=13points
4. A history of significant heart failure (New York Heart Association class III and IV)
5. Overt hepatic encephalopathy,
6. Prehepatic portal hypertension
7. Malignancy (including hepatocellular carcinoma) or a concomitant disease with reduced life expectancy
8. Uncontrolled infection and sepsis
9. Previous treatment to prevent rebleeding with a portosystemic shunt,TIPS or with pharmacological therapy with non-selective beta blockers and endoscopic variceal ligation
10. Pregnancy or lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-07-09 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause rebleeding or all-cause death | 3 years
  Cumulative incidence of all-cause rebleeding or all-cause death

SECONDARY OUTCOMES:
Portal vein recanalization | 3 years
  Incidence of portal vein recanalization
Other decompensations of portal hypertension | 3 years
  defined as ascites, spontaneous bacterial peritonitis, and hepatorenal syndrome
adverse events of treatment | 3 years
  Incidence of adverse events of treatment
Quality of life | 3 years
  quality of life assessed by the SF-36 health survey
Overall survival | 3 years
  Overall survival rate
Hepatocellular Carcinoma | 3 years
  Incidence of Hepatocellular Carcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Guohong Han, MD, Principal Investigator — Xi'an International Medical Center Hospital
Locations (8):
- China (8):
  - the First Affiliated Hospital, Air Force Medical University, Xi'an, Shaanxi
  - Xi'an International Medical Center Hospital, Xi'an, Shaanxi
  - Nanfang Hospital Affiliated to Southern Medical Univers, Guangzhou
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou
  - Provincial Hospital Affiliated to Shandong University, Jinan
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Affiliated Drum Tower Hospital of Nanjing University Medical School, Nanjing
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi

REFERENCES:
- [Background] Han G, Qi X, He C, Yin Z, Wang J, Xia J, Yang Z, Bai M, Meng X, Niu J, Wu K, Fan D. Transjugular intrahepatic portosystemic shunt for portal vein thrombosis with symptomatic portal hypertension in liver cirrhosis. J Hepatol. 2011 Jan;54(1):78-88. doi: 10.1016/j.jhep.2010.06.029. Epub 2010 Aug 27. PMID 20932597
- [Background] Lv Y, He C, Wang Z, Guo W, Wang J, Bai W, Zhang L, Wang Q, Liu H, Luo B, Niu J, Li K, Tie J, Yin Z, Fan D, Han G. Association of Nonmalignant Portal Vein Thrombosis and Outcomes after Transjugular Intrahepatic Portosystemic Shunt in Patients with Cirrhosis. Radiology. 2017 Dec;285(3):999-1010. doi: 10.1148/radiol.2017162266. Epub 2017 Jul 5. PMID 28682164